CLINICAL TRIAL: NCT05402319
Title: Comparison of Systemic (Mono-/Combination Therapies) and Topical Antibiotic Treatments Against Recurrent Urinary Tract Infections (RUTI) Caused by Multidrug Resistant Bacteria in Catheterized Patients
Brief Title: Comparison of Three Different Antibiotic Treatments Against Recurrent Urinary Tract Infections in Catheterized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Zhijun Song, Chief Physician, Associate Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Projekt-ID: S-20190083G CSF
Record Dates: First submitted 2022-05-16; First posted 2022-06-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Urinary Tract Infections; Chronic Urinary-catheter-carrier; Biofilm Infection; Antibiotic Treatment; Replacement of Urinary Catheter
Keywords: chronic urinary-catheter-carrier; recurrent urinary tract infection; biofilm infections; multidrug-resistant bacteria; antibiotic monotherapy; combination therapy; bladder lavage; urinary catheter replacement
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly into 3 individual groups: (1) systemic antibiotic monotherapy; (2) systemic antibiotic combination therapy; and (3) bladder antibiotic lavage (topical therapy).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be 150 patients involve in the study. The investigators have prepared 150 paper balls with numbers for the lottery. If the patient meets the inclusion criteria, the patient will be allowed to read the written instructions for invitation to participate in the study. The doctors and nurses will answer questions from patients. A signature is required if the patient agrees to participate in the study. The patient will then be allowed to draw a ball of paper, and the nurse or doctor will register the corresponding number in the computer. Patients 1-50 will be the first group, 51-100 the second group, and 101-150 the third group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antibiotic monotherapy (Experimental): Single antibiotic is given intravenously or orally (systemically).
  Interventions: Combination Product: Antibiotic combination therapy
- Antibiotic combination therapy (Experimental): At least two different antibiotics are given intravenously or orally.
  Interventions: Combination Product: Antibiotic combination therapy
- Topical antibiotic therapy (Experimental): Single antibiotic bladder irrigation.
  Interventions: Combination Product: Antibiotic combination therapy

INTERVENTIONS:
Combination Product: Antibiotic combination therapy — Anti-infective treatment with at least two different types of sensitive antibiotics.
  Other Names: Systemic versus topical antibiotic therapies

SUMMARY:
Recurrent urinary tract infections (UTI) in the patients chronically catheterized are serious challenges clinically. The pathogens are often multidrug-resistant bacteria and such UTIs are actually biofilm infections. Currently standard antibiotic treatment against UTI in Denmark is sensitive antibiotic monotherapy. Theoretically antibiotic monotherapy is not a good treatment against biofilm infections. In the patients with impaired renal functions, both i.v. and p.o. antibiotic treatments function poor. Therefore, bladder lavage might help. In the study, the participants will be randomly divided into three groups (monotherapy, combination and bladder lavage). The investigators will evaluate the results and find a better treatment based on the clinical evidences, which might benefit the patients.

DETAILED DESCRIPTION:
Multidrug resistant bacterial infections are serious challenges that human beings are facing. Recurrent urinary tract infections (UTI) in the patients chronically catheterized is one of the examples. Urinary catheterization not only impair the urinary tract self-clean mechanism, but also provide the urinary pathogens an ideal surface to form bacterial biofilms, which have been demonstrated in vivo and in vitro impossible to be removed by only antibiotic treatments. Repeated antibiotic treatments could not help to remove urinary biofilm infections, but induction of antibiotic resistance.

Currently treatment against recurrent UTI in urinary catheterized patients includes antibiotic treatment and replacement of urinary catheter. Antibiotic treatment aims to remove the planktonic bacteria, control clinical symptoms and localize the infection in urinary tract, which will help to limit the bacteria in the catheter biofilm and benefit the replacement of the infected catheter. At present, standard antibiotic treatment against UTI in catheter carriers is sensitive antibiotic monotherapy according to the Danish guidelines on the use of antibiotics in the website "https://pro.medicin.dk/". However, these kinds of UTIs are usually biofilm infections, especially the urinary pathogen are quite often multiple-resistant. Therefore, some of the hospitals prefer combination antibiotic treatments according to the results from biofilm in vivo and in vitro researches. There are currently always arguments regarding monotherapy and combination antibiotic treatments. The investigators intends to observe and compare both treatments and try to clarify their respective advantages and disadvantages, which will benefit the clinical treatments and control of the antibiotic resistance in future. In addition, some of the patients have poor renal function, which reduce significantly the antibiotic concentration in urine. In such situation, bladder-antibiotic lavage might help. In the study, the patients will be randomly divided into three groups (monotherapy, combination and bladder lavage). The investigators will evaluate the results and find a better treatment based on the clinical evidences, which might benefit the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who have long-term urinary catheter in situ with recurrent UTI and are admitted or referred to an ambulatory due to acute episode of UTI (acute local symptoms include pyuria or urine stick positive, suprapubic pain or tenderness, costovertebral angle pain or tenderness, catheter obstruction, or acute hematuria) or urosepsis (If a bacteriuric patient has positive blood culture with fever, leukocytosis and high C-reaction protein, and the cultured bacteria in urine and blood are consistent, urosepsis is diagnosed) will be included to the project.

Exclusion Criteria:

* Patients with nephrostomy catheters, J-J catheter, bricker bladder or urinary stones will be excluded from the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Infection control | 3 days
  Local UTI symptoms (cloudy urine, hematuria, smelly urine, discomfort or pain in the lower abdomen or pubic symphysis) were significantly reduced or disappeared.
Infection control | Less than 3 days
  Higher body temperature (more than 37.5 degrees) recover to normal (between 36 - 37 degrees).
Infection control | Less than or equal to 5 days
  Blood leukocyte count reduced from more than 8,800 × 109/L (dominated by neutrophils) to between 4,000 to 8,800 x 109/L.
Infection control | Less than or equal to 5 days
  C-reactive protein (CRP) reduced from significantly higher than 10 mg/L to less than 10 mg/L.
Infection control | Less than or equal to 5 days
  Estimated glomerular filtration rate (eGFR) recovered from less than 60 mL/min/1,73 m2 to equal to 60 or higher.

SECONDARY OUTCOMES:
UTI recurrence expectation | One month
  Significant less UTI recurrence.